CLINICAL TRIAL: NCT00421018
Title: Optimization of the Anti-Inflammatory Treatment of Asthma Patients Through Exhaled NO Measurements for Increased Asthma-Related Quality of Life in Primary Health Care (NOAK)
Brief Title: Optimization of Asthma Treatment Through Exhaled NO for Increased Asthma-Related Quality of Life (NOAK)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); Aerocrine AB (Industry); Phadia AB (Unknown); Meda AB (Unknown); The Swedish Research Council (Other Government); Swedish Council for Working Life and Social Research (Other); Merck Sharp & Dohme LLC (Industry); Uppsala University (Other)
Responsible Party: Kjell Alving/ Professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20050166
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Allergic Asthma
Keywords: Asthma; Allergy; Cytokines; Glucocorticoids; Inflammation; Nitric Oxide (NO); Quality of Life; Self-Rated Health; Stress
MeSH Terms: conditions — Asthma; Hypersensitivity; Inflammation | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Symptom-guided group (Sham Comparator): Anti-inflammatory treatment is guided conventionally according to symptoms and beta-2-agonist use.
  Interventions: Drug: Single corticosteroid inhalers and Singulair
- FeNO-guided group (Active Comparator): Anti-inflammatory treatment is guided according to the level of exhaled nitric oxide
  Interventions: Drug: Single corticosteroid inhalers and Singulair

INTERVENTIONS:
Drug: Single corticosteroid inhalers and Singulair — Treatment steps according to preset algorithm

SUMMARY:
The purpose of this study is to determine whether use of exhaled NO (nitric oxide) to regulate the anti-inflammatory treatment leads to increased asthma-related quality of life in patients with allergic asthma

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64
* Clinical diagnosis of Asthma
* Glucocorticoid treatment > 6 months.
* Verified Allergy
* Read and speak Swedish

Exclusion Criteria:

* Smoking
* Current regular treatment with long-acting beta2-agonist
* Treatment with Singulair only or in combination with glucocorticoids
* Taking part in other research study
* Pregnancy or breast-feeding
* Unstable Asthma

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 187 (Actual)
Dates: Start 2006-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Mini-AQLQ (Asthma-Related Quality of Life) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kjell Alving, PhD, Principal Investigator — Uppsala University
Locations (1):
- Runby Primary Health Care Center, Upplands Vasby, Sweden